CLINICAL TRIAL: NCT06196346
Title: Inter-Brain Synchrony in Psychotherapy for Depression
Acronym: IBSPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Society for the Advancement of Psychotherapy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 047/21
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: Synchrony; fNIRS; Imaging; Psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study was designed to examine changes in inter-brain synchrony over the course of standard psychotherapy, and not treatment effectiveness. As such, a single group design was deemed adequate.
Masking Description: There was no assignment to different groups and as a result, no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Main group (Experimental): The group underwent 16 sessions of supportive-expressive psychotherapy (Luborsky et al., 1995)
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — see group description

SUMMARY:
The study aims to examine inter-brain synchrony between patients and therapists over the course of psychotherapy. Twenty patients will undergo a 16-session course of psychotherapy for major depressive disorder. The protocol used will be supportive-expressive psychotherapy (see Luborsky et al., 1995). Participants will also undergo Hamilton depression interviews a week before treatment, before every session and a week after treatment. functional near-infrared spectroscopy (fNIRS) imaging will be used to record brain activity during every other session (sessions 1, 3, 5, 7, 9, 11, 13, 15) as well as during interviews at baseline, on session 8 and at followup. Saliva samples will be collected during the same sessions to measure hormone and cytokine levels during the same sessions. Participants completed questionnaires before and after the study, and before and after each session.

The researchers hypothesized that synchrony will gradually increase over the psychotherapy sessions, and that synchrony in the pre-treatment interview will be lower than in the post-treatment interview.

DETAILED DESCRIPTION:
This study centers on a 16-session supportive-expressive treatment protocol for major depression (Luborsky et al., 1995).

The study will last 18 weeks. On weeks 1 and 18 participants will come in to a screening interview preformed by a research assistant. On weeks 2-17 participants will come in to therapy meetings, according to the aforementioned protocol. Every week prior to screening / treatment participants will also undergo a Hamilton depression interview. On weeks 1,2,4,6,8,9,10,12,14,16,18 the researchers will also perform functional near-infrared spectroscopy (fNIRS) imaging and take saliva samples (on weeks 1,9, and 18 - during the Hamilton interview. On other weeks - during treatment). Participants, interviewers (when interviews were assessed) and therapists (when treatment was assessed) underwent fNIRS imaging and provided saliva samples to measure Oxytocin, Cortisol and Cytokine levels. Samples will be tested for levels and subsequently destroyed.

All therapists will be licensed psychologists, and will performing a brief version of Supportive-Expressive therapy (Luborsky et al., 1995). Therapists have all undergone specific training in Supportive-Expressive therapy before being involved in the study. They will also have a group supervision meeting once every two weeks with a therapist who is highly experienced in Supportive-Expressive therapy.

Participants will also complete self-report questionnaires - for some of the questionnaires they may be given the option to complete them online outside of the weekly meeting itself.

ELIGIBILITY:
Inclusion Criteria:

* : (a) meeting MDD diagnostic criteria using the DIAMOND structured clinical interviews for DSM-V, and scoring more than 8 on the 17-item Hamilton Rating Scale for Depression (HRSD; Hamilton, 1967) at two evaluations, one week apart; (b) if on medication, patients' dosage must be stable for at least three months before the study, and they must be willing to maintain stable dosage for the duration of treatment; (c) age between 18 and 70; (d) Hebrew language fluency; (e) provision of written informed consent.

Exclusion Criteria:

* (a) HRSD suicide item > 2; (b) current substance abuse disorders; (c) current or past schizophrenia or psychosis, bipolar disorder, or severe eating disorder requiring medical monitoring; (d) history of organic mental disease (but having ADHD will not disqualify participants); (e) currently in psychotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression | Weeks 1,18
  A t-test will examine whether participants' scores on the Hamilton depression interview (Hamilton, 1967) have been reduced.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
Numerical questionnaire data, hormone levels and fNIRS recordings will be made available to other researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication
Access Criteria: Open access

REFERENCES:
- [Background] Luborsky, L., Mark, D., Hole, A. V., Popp, C., Goldsmith, B., & Cacciola, J. (1995). Supportive-expressive dynamic psychotherapy of depression: A time-limited version. In J. P. Barber & P. Crits-Christoph (Eds.), Dynamic therapies for psychiatric disorders (Axis I) (pp. 13-42). Basic Books.
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235